CLINICAL TRIAL: NCT00769834
Title: Incidence and Causes of Disc Edema in Patients With Chronic Kidney Disease
Brief Title: Disc Edema in Patients With Chronic Kidney Disease
Status: Withdrawn | Type: Observational
Why Stopped: All investigators have moved to different oranizations
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Sachin Kedar, Faculty, University of Nebraska
Other Study IDs: 2008-0019
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; chronic renal insufficiency; uremia; disc edema; papilledema; idiopathic intracranial hypertension; pseudotumor cerebri
MeSH Terms: conditions — Renal Insufficiency, Chronic; Uremia; Papilledema; Pseudotumor Cerebri

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CKD: The cohort comprises of patients who are diagnosed to have chronic kidney disease as defined by the K/DOQI Clinical Practice Guidelines for Chronic Kidney Disease-2002.

SUMMARY:
Papilledema is defined as swelling of the optic nerves often due to increased intracranial pressure. When present, it often indicates life-threatening lesions of the brain such as tumors, abscesses, meningitis, encephalitis, venous sinus obstruction or intracranial hemorrhage. A similar clinical picture can also be caused by other conditions such as malignant hypertension, diabetic papillopathy and uremia. When the intracranial pressure is elevated in the absence of any known cause then it is called Idiopathic Intracranial Hypertension (IIH). Untreated papilledema can cause progressive optic nerve damage and blindness.

Patients with chronic kidney disease have a number of co-morbidities and thus are at an increased risk for developing papilledema. Although clinicians have observed that patients with kidney diseases have increased incidence of papilledema (unpublished data by Corbett et al), there have been no studies on this subject to date. We believe that a higher incidence of papilledema is found in patients with kidney diseases and this study could provide evidence to suggest routine ophthalmic screening in this patient group.

Hypothesis: The prevalence of optic disc swelling is increased in patients with chronic kidney disease.

Purpose: To establish the prevalence of disc edema in patients with chronic kidney disease.

DETAILED DESCRIPTION:
The craniospinal cavity is enclosed by a rigid, non-compressible bone and thus has a constant volume. It is filled with soft tissue (brain, spinal cord and connective tissue), cerebrospinal fluid (CSF) and circulating blood. Intracranial pressure (ICP) is the pressure of the fluid that bathes the brain and the spinal cord. The ICP is regulated by a fine balance between the production and absorption of CSF. Any disturbance in the volumes of the contents of the rigid craniospinal cavity will cause an alteration of the ICP. Intracranial pressure can be elevated from a number of disease processes such as space occupying lesions, abnormalities of the production and absorption of the CSF and abnormalities of the circulation such as venous obstruction.

Raised ICP will symptomatically manifest as headache, vomiting, tinnitus and diplopia in addition to neurologic symptoms related to the lesion location and type. The increased ICP can be transmitted to the optic nerves causing papilledema, defined as swelling of the optic nerve head (papilla) secondary to raised ICP. Swelling of the optic nerves in the absence of raised ICP is termed disc edema (Parsons JH, Miller NR). Causes of disc edema are extensive and include ischemic optic neuropathy, malignant hypertension, diabetic papillopathy, uremia, intracranial hypotension (CSF leak).

Papilledema is considered a medical emergency and is investigated by means of neuroimaging (to evaluate intracranial lesions) and lumbar puncture (to evaluate the opening pressure and CSF contents). A diagnosis of Idiopathic Intracranial Hypertension (IIH) is made when there is elevated ICP in the absence of clinical, laboratory or radiological evidence of any known cause of raised ICP.

The most feared complication of untreated papilledema is progressive optic nerve atrophy resulting in vision loss. Early recognition, investigation and treatment of papilledema and its causes can prevent blindness.

Patients with chronic kidney diseases have a number of risk factors which predispose them to the development of disc edema. Medical comorbidities such as hypertension and diabetes mellitus increase their risk for optic nerve head diseases such as ischemic optic neuropathy and diabetic papillopathy. Malignant hypertension, uremia and dialysis dysequilibrium syndrome also are known to cause papilledema.

There are no studies in the English literature to date, on disc edema in patients with kidney diseases. However, neuroophthalmologists have clinically observed that patients with chronic kidney diseases appear to have an increased incidence of optic nerve swelling (Corbett JJ, unpublished data). A study looking at optic nerve edema in this group of patients is overdue and may determine additional guidelines in the management of patients with chronic kidney diseases.

The patients enrolled in the study will undergo an optic nerve head examination by ophthalmoscopy to identify patients with disc edema. If disc edema is detected on the screening examination, the patients will be referred to the Neuroophthalmology service for evaluation and investigations to determine the further management. The results of the neuroophthalmologic workup for patients with disc edema will be reviewed to ascertain the etiology of disc edema.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have been identified to have kidney disease (as defined by the K/DOQI Clinical Practice Guidelines for Chronic Kidney Disease-2002)

Exclusion Criteria:

* Patients with renal transplantation
* Patients who are less than 18 years of age
* Patients who are unable to provide an informed consent to participate in the study.
* Chronic Steroid use greater than or equal to 3 months within the last 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will be drawn from the population of patients with chronic kidney diseases attending the kidney disease clinics and the hemodialysis units at the University of Mississippi Medical Center and the Jackson Medical Mall
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
disc edema | 0 days

SECONDARY OUTCOMES:
ophthalmoscopic diagnosis | 0 days
neurologic diagnosis | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: SACHIN KEDAR, M.D, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Im L, Atabay C, Eller AW. Papilledema associated with dialysis disequilibrium syndrome. Semin Ophthalmol. 2007 Jul-Sep;22(3):133-5. doi: 10.1080/08820530701421585. PMID 17763231
- [Background] Chang S, Masaryk TJ, Lee MS. Optic nerve edema: complication of peripheral hemodialysis shunt. Semin Ophthalmol. 2004 Sep-Dec;19(3-4):88-90. doi: 10.1080/08820530490882319. PMID 15590543
- [Background] Dogulu CF, Tsilou E, Rubin B, Fitzgibbon EJ, Kaiser-Kupper MI, Rennert OM, Gahl WA. Idiopathic intracranial hypertension in cystinosis. J Pediatr. 2004 Nov;145(5):673-8. doi: 10.1016/j.jpeds.2004.06.080. PMID 15520772
- [Background] Khositseth S, Chavers BM, Czapansky-Beilman D, Mauer M. Idiopathic intracranial hypertension immediately after kidney transplantation in a pediatric recipient. Pediatr Nephrol. 2004 Dec;19(12):1416-7. doi: 10.1007/s00467-004-1616-8. PMID 15378420
- [Background] Francis PJ, Haywood S, Rigden S, Calver DM, Clark G. Benign intracranial hypertension in children following renal transplantation. Pediatr Nephrol. 2003 Dec;18(12):1265-9. doi: 10.1007/s00467-003-1274-2. Epub 2003 Oct 30. PMID 14586682
- [Background] Obeid T, Awada A, Huraib S, Quadri K, Abu-Romeh S. Pseudotumor cerebri in renal transplant recipients: a diagnostic challenge. J Nephrol. 1997 Sep-Oct;10(5):258-60. PMID 9364317
- [Background] Koller EA, Stadel BV, Malozowski SN. Papilledema in 15 renally compromised patients treated with growth hormone. Pediatr Nephrol. 1997 Aug;11(4):451-4. doi: 10.1007/s004670050315. PMID 9260244
- [Background] Katz B. Disk edema subsequent to renal transplantation. Surv Ophthalmol. 1997 Jan-Feb;41(4):315-20. doi: 10.1016/s0039-6257(96)00006-9. PMID 9104768
- [Background] Sheth KJ, Kivlin JD, Leichter HE, Pan CG, Multauf C. Pseudotumor cerebri with vision impairment in two children with renal transplantation. Pediatr Nephrol. 1994 Feb;8(1):91-3. doi: 10.1007/BF00868279. PMID 8142239
- [Background] Chang D, Nagamoto G, Smith WE. Benign intracranial hypertension and chronic renal failure. Cleve Clin J Med. 1992 Jul-Aug;59(4):419-22. doi: 10.3949/ccjm.59.4.419. PMID 1525975
- [Background] Niutta A, Scorcia G, Princi P, Palombi E, Perilli R, Mannino G, Balacco Gabrieli C. Visual disturbances associated with primary empty sella syndrome in patients with chronic renal failure. Ann Ophthalmol. 1992 Feb;24(2):56-63. PMID 1562126
- [Background] Hamed LM, Winward KE, Glaser JS, Schatz NJ. Optic neuropathy in uremia. Am J Ophthalmol. 1989 Jul 15;108(1):30-5. doi: 10.1016/s0002-9394(14)73256-8. PMID 2750832
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Guy J, Johnston PK, Corbett JJ, Day AL, Glaser JS. Treatment of visual loss in pseudotumor cerebri associated with uremia. Neurology. 1990 Jan;40(1):28-32. doi: 10.1212/wnl.40.1.28. PMID 2296378
- [Background] Taban M, Taban M, Lee MS, Smith SD, Heyka R, Kosmorsky GS. Prevalence of optic nerve edema in patients on peripheral hemodialysis. Ophthalmology. 2007 Aug;114(8):1580-3. doi: 10.1016/j.ophtha.2006.10.060. Epub 2007 Mar 21. PMID 17368544